CLINICAL TRIAL: NCT01378520
Title: The Effect of Ketoconazole on Breathlessness During Resistive Load Breathing in Patients With Chronic Obstructive Pulmonary Disease
Brief Title: Effect of Ketoconazole on Breathlessness
Acronym: KetoRLB
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Dartmouth-Hitchcock Medical Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CPHS22775
Record Dates: First submitted 2011-06-16; First posted 2011-06-22 (Estimated); Results first posted 2013-11-14 (Estimated); Last update posted 2018-06-01 (Actual); Status verified 2018-05

CONDITIONS: Chronic Obstructive Pulmonary Disease
Keywords: breathlessness; resistive load breathing; beta-endorphins
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive; Dyspnea | interventions — Ketoconazole; Antifungal Agents

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- ketoconazole (Experimental): 600 mg ketoconazole
  Interventions: Drug: ketoconazole
- inert powder (Placebo Comparator): inert powder in capsule
  Interventions: Drug: inert powder

INTERVENTIONS:
Drug: ketoconazole — 600 mg capsule oral once
  Other Names: oral antifungal
  Arms: ketoconazole
Drug: inert powder — oral once
  Other Names: oral placebo
  Arms: inert powder

SUMMARY:
Beta-endorphins, which are naturally occurring narcotic substances, have been shown to alter the perception of breathlessness. Oral ketoconazole, an antifungal antibiotic, increases blood levels of beta-endorphins. The study hypothesis is that oral ketoconazole will reduce ratings of breathlessness induced by resistive breathing loads.

DETAILED DESCRIPTION:
Beta-endorphins are naturally occurring narcotic substances (like morphine) that are released by the brain under stressful conditions, such as exercise and when breathing through a resistive load (a tube containing fine wire mesh). In one study of 8 patients with coronary artery disease, ketoconazole, an oral medication used to treat fungal infections, was administered (1,200 mg at 12 midnight and 600 mg at 6 am) and increased blood levels of beta-endorphins five fold. In a recent study performed at Dartmouth-Hitchcock Medical Center, we found that ketoconazole increased blood levels of beta-endorphins in all eight patients with chronic obstructive pulmonary disease (COPD). Mean values increased by 2.5 times at four hours compared with baseline values (p = 0.0078). Based on this significant response, we propose to study the effect of ketoconazole on patients' perception of breathlessness induced by resistive breathing loads in a randomized clinical trial. The hypothesis of the study is that ketoconazole will reduce ratings of breathlessness as mediated by the increased levels of beta-endorphins.

ELIGIBILITY:
Inclusion Criteria:

* 50 years of age or older;
* diagnosis of COPD;
* current or former smoker of at least 10 pack-years;
* post-bronchodilator FEV1 greater than or equal to 30% predicted and less than or equal to 80% predicted; post-bronchodilator ratio < 70%

Exclusion Criteria:

* any concomitant disease that might interfere with study procedures;
* use of a drug that may cause a possible drug interaction with ketoconazole

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2011-06; Primary Completion 2012-02 (Actual); Study Completion 2012-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Donald A Mahler, MD, Principal Investigator — Dartmouth-Hitchcock Medical Center
Locations (1):
- Dartmouth-Hitchcock Medical Center, Lebanon, New Hampshire, United States

REFERENCES:
- [Background] Gifford AH, Mahler DA, Waterman LA, Ward J, Kraemer WJ, Kupchak BR, Baird JC. Neuromodulatory effect of endogenous opioids on the intensity and unpleasantness of breathlessness during resistive load breathing in COPD. COPD. 2011 Jun;8(3):160-6. doi: 10.3109/15412555.2011.560132. Epub 2011 Apr 22. PMID 21513438
- [Derived] Mahler DA, Gifford AH, Waterman LA, Ward J, Kraemer WJ, Kupchak BR, Harver A. Effect of increased blood levels of beta-endorphin on perception of breathlessness. Chest. 2013 May;143(5):1378-1385. doi: 10.1378/chest.12-1541. PMID 23715032

RESULTS

PARTICIPANT FLOW:
Recruitment Details: June 2011 - January 2012; medical center
Pre-assignment Details: 23 subjects recruited; 1 excluded (did not meet inclusion/exclusion criteria); 2 withdrawn prior to randomization (1 could not tolerate breathing through the initial inspiratory resistance (15 cm H 2 O/L/s); 1 gave ratings of breathlessness of < 50 mm on the VAS for the highest resistance (50 cm H2O/L/s))
Groups:
- First Ketoconazole, Then Inert Powder: Ketoconzaole (600 mg taken orally) in first intervention period and inert powder (in capsule taken orally) in second intervention period.
- First Inert Powder, Then Ketoconazole: Inert powder (in capsule taken orally) in first intervention period and Ketoconzaole (600 mg taken orally) in second intervention period.
Period: First Intervention (Day 2-3)
Arm/Group | First Ketoconazole, Then Inert Powder | First Inert Powder, Then Ketoconazole
Started | 10 | 10
Completed | 10 | 10
Not Completed | 0 | 0
Period: Second Intervention (Day 4-6)
Arm/Group | First Ketoconazole, Then Inert Powder | First Inert Powder, Then Ketoconazole
Started | 10 | 10
Completed | 10 | 10
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Entire Study Population: Includes groups randomized to receive Ketoconazole first and inert powder first.
Arm/Group | Entire Study Population
Number analyzed (Participants) | 20
Age, Continuous [Mean (Standard Deviation); unit: years] | 69.6 (6.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 10
  Male | 10
Region of Enrollment [Number; unit: participants]
  United States | 20

OUTCOME MEASURES:

1. Primary Outcome: Unpleasantness of Breathlessness
Description: The average of all ratings for the unpleasantness of breathlessness at equivalent times for each subject during Resistive Load Breathing (RLB). For example, if 1 subject provided 6 ratings during 6 minutes of RLB with Ketoconazole and 10 ratings during 10 minutes of RLB with inert powder, then ratings for unpleasantness through 6 minutes were used for analysis for that patient. This approach was used for all subjects to yield a total of 252 ratings for Ketoconazole and for inert powder.
  Subject rating of intensity of unpleasantness was obtained during RLB on a 100 mm Visual Analog Scale anchored at the bottom by "No Unpleasantness" and at the top by "Greatest Unpleasantness".
Time Frame: At 1 minute intervals during Resistive Load Breathing at Period 1 (Day 3 or 4) and Period 2 (Day 5, 6 or 7)
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- Ketoconazole: Ketoconazole (600 mg given orally)
- Inert Powder: Inert powder (in capsule taken orally)
Arm/Group | Ketoconazole | Inert Powder
Number analyzed (Participants) | 20 | 20
units on a scale | 72.5 (23.8) | 72.6 (23.5)

2. Primary Outcome: Intensity of Breathlessness
Description: The average of all ratings for the intensity of breathlessness at equivalent times for each subject during Resistive Load Breathing (RLB). For example, if 1 subject provided 6 ratings during 6 minutes of RLB with Ketoconazole and 10 ratings during 10 minutes of RLB with inert powder, then ratings for intensity through 6 minutes were used for analysis for that patient. This approach was used for all subjects to yield a total of 252 ratings for Ketoconazole and for inert powder.
  Subject rating of intensity of breathlessness was obtained at 1 minute intervals during RLB on a 100 mm Visual Analog Scale anchored at the bottom by "No Intensity" and at the top by "Greatest Intensity".
Time Frame: At 1 minute intervals during Resistive Load Breathing at Period 1 (Day 3 or 4) and Period 2 (Day 5, 6 or 7)
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Ketoconazole | Inert Powder
Number analyzed (Participants) | 20 | 20
units on a scale | 77.6 (22.3) | 78.2 (21.4)

3. Secondary Outcome: Change in Level of B-endorphin Immunoreactivity
Description: Change between pre-treatment and post treatment serum levels of beta-endorphin immunoreactivity measured in pmol/L
Time Frame: At the end of resistance load breathing (4.5 hours after receiving the test article)
Measure: Mean (Standard Deviation); unit: pmol/L
Arm/Group | Ketoconazole | Inert Powder
Number analyzed (Participants) | 20 | 20
pmol/L | 153.9 (18.0) | 93.9 (7.9)

ADVERSE EVENTS:
Groups:
- Ketoconazole: Ketoconazole(600 mg taken orally)
Arm/Group | Ketoconazole | Inert Powder
Serious Adverse Events (participants affected / at risk) | 0/10 | 0/10
Other Adverse Events (participants affected / at risk) | 0/10 | 0/10

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No